CLINICAL TRIAL: NCT02540226
Title: The Effect of Topical and Intravenous Tranexamic Acid (TXA) on Thrombogenic Markers in Patients Undergoing Total Knee Replacement
Brief Title: Effect of Topical and Intravenous Tranexamic Acid (TXA) on Thrombogenic Markers in Patients Undergoing Knee Replacement
Acronym: TXA Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-210
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Tranexamic Acid; Total Knee Arthroplasty; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous tranexamic acid (Active Comparator): Patients will receive 1g tranexamic acid in 100mL solution intravenously in the operating room before inflation of the tourniquet. They will again receive the same IV solution in the post-anesthesia care unit, approximately 3 hours after the first solution was given. They will also receive a 75cc topical saline solution approximately 5 minutes before the tourniquet is released.
  Interventions: Drug: Intravenous tranexamic acid; Drug: Topical saline
- Topical tranexamic acid (Experimental): Patients will receive 3g tranexamic acid in 75mL solution topically in the operating room, approximately 5 minutes before the tourniquet is released. It will sit for 5 minutes before the solution is suctioned off by the surgeon. They will also receive 2 intravenous saline solutions: one in the operating room before inflation of the tourniquet, and one in the post-anesthesia care unit 3 hours after the first solution was given.
  Interventions: Drug: Topical tranexamic acid; Drug: Intravenous saline

INTERVENTIONS:
Drug: Intravenous tranexamic acid
  Arms: Intravenous tranexamic acid
Drug: Topical tranexamic acid
  Arms: Topical tranexamic acid
Drug: Intravenous saline
  Arms: Topical tranexamic acid
Drug: Topical saline
  Arms: Intravenous tranexamic acid

SUMMARY:
Tranexamic acid (TXA) is a drug that is being used more frequently at the Hospital for Special Surgery to lessen the amount of blood loss after total knee replacement (TKR). It is an anti-fibrinolytic agent, which means that it promotes the formation of blood clots. TXA can be given either intravenously or topically (placed directly on the open wound) before wound closure. Patients with certain medical conditions have been found to have a high risk of thrombosis after being given intravenous TXA, which may lead to serious complications. However, to date, no high-risk patients have been identified for use of topical TXA. This study will look at thrombogenic markers (proteins found in blood that promote clot formation) after TXA is given either intravenously or topically. If the effect on these markers is similar between intravenous and topical use of TXA, then the safety of topical TXA should be questioned. Of note, these markers have never been measured after TXA has been given topically. As a result, this information would be important for the medical community.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary unilateral total knee replacement with a participating surgeon
* Patients aged 18-80

Exclusion Criteria:

* All patients on steroid therapy regardless of dose, duration, or treatment or those requiring stress-dose steroids preoperatively
* Patients who will require postoperative use of Coumadin, Xarelto, or Plavix
* Use of non-steroidal anti-inflammatory drugs (NSAIDs) within 1 week of surgery
* Hypersensitivity to tranexamic acid
* Renal dysfunction (Creatinine clearance < 40 ml/min)
* Hepatic dysfunction (AST or ALT 2x upper limit of normal)
* Cardiac exclusions: coronary stent, history of myocardial infarction, positive stress test, atrial fibrillation, advanced coronary artery disease
* Advanced chronic obstructive pulmonary disease or advanced interstitial lung disease
* History of venous thromboembolism
* Hypercoagulability (e.g. antiphospholipid syndrome, genetic hypercoagulability with or without prior venous thromboembolism)
* History of stroke or transient ischemic attack

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kethy Jules-Elysee, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Tranexamic Acid: Patients will receive 1g tranexamic acid in 100mL solution intravenously in the operating room before inflation of the tourniquet. They will again receive the same IV solution in the post-anesthesia care unit, approximately 3 hours after the first solution was given. They will also receive a 75cc topical saline solution approximately 5 minutes before the tourniquet is released.
  Intravenous tranexamic acid
  Topical saline
- Topical Tranexamic Acid: Patients will receive 3g tranexamic acid in 75mL solution topically in the operating room, approximately 5 minutes before the tourniquet is released. It will sit for 5 minutes before the solution is suctioned off by the surgeon. They will also receive 2 intravenous saline solutions: one in the operating room before inflation of the tourniquet, and one in the post-anesthesia care unit 3 hours after the first solution was given.
  Topical tranexamic acid
  Intravenous saline
Period: Overall Study
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Started | 33 | 33
Completed | 31 | 32
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (8.4) | 65.0 (6.9) | 65.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 32
  Male | 11 | 20 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 31 | 28 | 59
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (7.1) | 31.1 (5.2) | 31.4 (6.2)
ASA Grade (II/III) [Count of Participants; unit: Participants] — ASA II -A patient with mild systemic disease; Mild diseases only without substantive functional limitations.
  ASA III- A patient with severe systemic disease; Substantive functional limitations; One or more moderate to severe diseases.
  Participants
    ASA II | 28 | 32 | 60
    ASA III | 3 | 0 | 3
Preoperative Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 135 (11) | 138 (11) | 136.4 (11.3)
Preoperative Hematocrit [Mean (Standard Deviation); unit: %] | 40.8 (3.2) | 41.0 (2.8) | 40.9 (3.0)
Preoperative Platelet count [Mean (Standard Deviation); unit: platelets/uL] | 241 (50) | 241 (60) | 241.0 (55.1)

OUTCOME MEASURES:

1. Primary Outcome: Levels of Plasmin Anti-plasmin (PAP) - Marker of Fibrinolysis
Description: Levels of PAP will be measured in peripheral blood and wound drainage at 4 hours after tourniquet release.
Time Frame: 4 hours after tourniquet release
Population: A wound drain was not inserted in all patients - hence why wound blood was not able to be collected 4 hours post tourniquet release.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 31 | 32
ug/L
  Systemic PAP blood level 4 HR post TQR | 117.8 (478.9) | 1280.7 (646.5)
  Wound PAP Blood Level 4 HR post TQR: number analyzed (Participants) | 26 | 31
  Wound PAP Blood Level 4 HR post TQR | 1032 (354.4) | 1041.2 (365.8)

2. Secondary Outcome: Levels of Prothrombin Fragment 1.2 (PF1.2) - Marker of Thrombin Generation
Description: Systemic PAP blood level measured at the following time points - Intraoperative - Before cementing, 1 hour after tourniquet release, 4 hours after tourniquet release
Time Frame: before cementing, 1 hour after tourniquet release, 4 hours after tourniquet release
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 31 | 32
pmol/L
  Intraoperative (before cemeting) | 400.2 (235.6) | 377.3 (218.4)
  1 hour after tourniquet release | 661 (243.5) | 636.2 (241.6)
  4 hour after tourniquet release | 812.9 (349.9) | 868.8 (336.2)

3. Secondary Outcome: Levels of Tranexamic Acid
Time Frame: Intraoperative (before cementing), 1 hour after tourniquet release (TQR), 4 hours after tourniquet release(TQR)
Population: Blood was collected from the A-Line or CostaVac Drain. If no drain was placed, the wound 4 hour post TQR blood could not be collected.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 31 | 32
mg/L
  Systemic Level - Intraoperative (before cemeting) | 31.0 (15.2) | 3.9 (13.1)
  Systemic Level - 1 Hour Post TQR | 19.9 (8.3) | 7.2 (7.4)
  Systemic Level - 4 Hour Post TQR | 27.4 (13.7) | 5.2 (8.8)
  Wound Level - Intraoperative (before cemeting) | 21.1 (11.2) | 2.2 (9.2)
  Wound Level - 4 Hour Post TQR: number analyzed (Participants) | 26 | 31
  Wound Level - 4 Hour Post TQR | 37.9 (16.1) | 31.4 (47.0)

4. Secondary Outcome: Calculated Postoperative Blood Loss
Time Frame: Duration of inpatient hospital stay (average of 3 days)
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 31 | 32
mL | 1237 [780 to 1456] | 1405 [1208 to 1700]

5. Secondary Outcome: Levels of Hemoglobin
Time Frame: 1 hour after tourniquet release, POD 1, POD 2
Population: The number in one or more rows differs from overall number analyzed because patients were either discharged early or there was a missing blood draw.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 31 | 32
g/dL
  1 hour after tourniquet release | 11.29 (1.21) | 11.41 (1.02)
  POD1: number analyzed (Participants) | 30 | 31
  POD1 | 11.12 (1.04) | 10.53 (0.13)
  POD2: number analyzed (Participants) | 30 | 32
  POD2 | 10.28 (1.19) | 9.94 (1.03)

6. Secondary Outcome: Levels of Hematocrit
Time Frame: 1 hour after tourniquet release, POD 1, POD 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: % of red blood cells in blood
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 31 | 32
% of red blood cells in blood
  1 hour after tourniquet release | 33.6 (3.6) | 33.8 (2.6)
  POD1: number analyzed (Participants) | 30 | 31
  POD1 | 35.6 (12) | 31.5 (4)
  POD2: number analyzed (Participants) | 30 | 32
  POD2 | 31 (3.5) | 29.8 (2.7)

7. Secondary Outcome: Constavac Blood Drainage
Description: A wound drain is connected to a Constavac system, which postoperatively collects, filters, and allows for reinfusion of the patient's own blood. Shed blood passes through an internal prefilter and is collected in a reservoir.
Time Frame: 4 hours after tourniquet release
Population: Some patients did not get a contavac drain put in hence the discrepancy in analysis population description.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 28 | 32
mL | 100 [90 to 185] | 170 [118 to 240]

8. Secondary Outcome: Incidence of Thrombosis (DVT/PE)
Time Frame: Postoperative day 14 (2 weeks after surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 31 | 32
Participants | 0 | 0

9. Secondary Outcome: Patients Who Had 1 Unit of Blood Transfusion Administered
Time Frame: Duration of inpatient hospital stay (average of 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 31 | 32
Participants | 1 | 1

10. Secondary Outcome: Time to Physical Therapy Discharge
Time Frame: During Hospital Stay
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 31 | 32
days | 1.9 [1.8 to 2.8] | 2.9 [2.0 to 3.0]

11. Secondary Outcome: Length of Hospital Stay
Time Frame: Length of Hospital Stay
Measure: Median (Full Range); unit: days
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 31 | 32
days | 2.3 [2.0 to 2.9] | 3.0 [2.5 to 3.2]

12. Secondary Outcome: Levels of IL-6 in Blood
Time Frame: Intraoperative, 1 hour post Tourniquet Release (TQR), 4 hour post Tourniquet Release (TQR)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 31 | 32
pg/mL
  Intraoperative (before cemeting) | 1.1 (0.9) | 3.9 (11.5)
  Systemic Level - 1 Hour Post TQR | 1.8 (1.2) | 5 (12.7)
  Systemic Level - 4 Hour Post TQR | 17.2 (14.9) | 25.6 (33.9)
  Wound Blood - Intraoperative (before cemeting) | 5.2 (7.6) | 6.7 (12.1)
  Wound Level - 4 Hour Post TQR | 5774.8 (4360.7) | 4497.6 (3325.5)

13. Secondary Outcome: Levels of Plasmin Anti-plasmin (PAP) - Marker of Fibrinolysis
Description: Levels of PAP will be measured in peripheral blood and wound drainage
Time Frame: Intraoperative, 1 hour post Tourniquet Release (TQR)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 31 | 32
mg/L
  Systemic Blood - Intraoperative (before cemeting) | 31.0 (15.2) | 3.9 (13.1)
  Systemic Level - 1 Hour Post TQR | 19.9 (8.3) | 7.2 (7.4)
  Wound Blood - Intraoperative | 21.1 (11.2) | 2.2 (9.2)

14. Secondary Outcome: Levels of Prothrombin Fragment 1.2 (PF1.2) - Marker of Thrombin Generation in Wound Blood
Description: The values for the wound blood levels are given as the count of patients who had a level above the threshold of >3600 pmol/L.
Time Frame: Intraoperative, 4 hour post Tourniquet Release (TQR)
Population: Blood samples could not be collected at the 4-hour post tourniquet release for some patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
Number analyzed (Participants) | 31 | 32
Participants
  Intraoperative (before cemeting) | 16 | 14
  4 hour after tourniquet release: number analyzed (Participants) | 28 | 32
  4 hour after tourniquet release | 13 | 11

ADVERSE EVENTS:
Time Frame: Adverse Events data was collected during the length of stay in the hospital which has an average of 3 days.
Arm/Group | Intravenous Tranexamic Acid | Topical Tranexamic Acid
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 0/31 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT02540226/Prot_SAP_000.pdf